CLINICAL TRIAL: NCT05479214
Title: Effect of Adding Metformin to Insulin in Uncontrolled Diabetic Patients During the 3rd Trimester of Pregnancy on Glycemic Control, Fetal and Neonatal Outcomes ,Randomized Controlled Trial
Brief Title: Effect of Adding Metformin to Insulin in Uncontrolled Diabetic Patients During the 3rd Trimester of Pregnancy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ayman Hany, MD, Associate Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: reda-metformin
Record Dates: First submitted 2022-06-26; First posted 2022-07-29 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Diabetes Mellitus Pregnancy
MeSH Terms: conditions — Diabetes, Gestational | interventions — Metformin; Insulin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin Group (Experimental): will include 75 patients who will be treated with metformin ( 1gm with the 2 main meals ) combined with insulin therapy
  Interventions: Drug: Metformin; Drug: Insulin
- Insulin alone group (Experimental): will include 75 patients who will be treated with insulin alone
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Metformin — 1gm tablet with the 2 main meals
  Arms: Metformin Group
Drug: Insulin — subcutaneous insulin daily administration

SUMMARY:
Background Diabetes mellitus (DM) is a significant contributor to adverse obstetric and perinatal outcome. There is now clear and unequivocal evidence that adverse pregnancy outcomes are strongly linked to maternal hyperglycemia, both in the peri-conception period and throughout gestation. Although strict glycemic control does improve outcomes, there is still a higher rate of complications in women with DM and poorer perinatal outcomes .

The incidence of type 2 diabetes is rising worldwide at a remarkable rate IDF When receiving large doses of insulin, patients complain of pain at the site of injection leading to compliance issues and poor glycemic control. This can be explained as when taking large doses of insulin it leads to alter absorption kinetics because very large doses are delivered to one site, resulting in a failure to reduce postprandial hyperglycemia, but with later hypoglycemia once the insulin is absorbed. This poor glycemic control in mothers with diabetes leads to an increased risk of severe respiratory distress syndrome, low Apgar scores, neonatal hypoglycemia and neonatal intensive care unit (NICU) admissions .

Infants of mothers with diabetes have high rates of being born large for gestational age (LGA) and macrosomic (>4 or 4.5 kg). Macrosomia is associated with increased rates of perinatal asphyxia, meconium aspiration, hypoglycemia, shoulder dystocia, brachial plexus injury, skeletal injuries, and fetal death .

Metformin is among the oldest and most well studied oral anti hyperglycemic agents. Its efficacy has been demonstrated both in the primary prevention of disease and secondary prevention of diabetes-related morbidity and mortality. Because of metformin's proven efficacy, low cost, and minimal side effect profile, it is largely recommended as the first line, initial monotherapy and as part of any combination therapy (included with insulin) for the treatment and prevention of type II diabetes .

Metformin produces euglycemia by reducing insulin resistance, improving insulin sensitivity, reducing hepatic gluconeogenesis, and increasing peripheral glucose uptake and utilization.

DETAILED DESCRIPTION:
Objectives To determine whether the addition of metformin to a standard regimen of insulin is more effective in glycemic control , fetal and neonatal outcome than conventional insulin alone in uncontrolled diabetic patients during the 3rd trimester of pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* • Diabetic pregnant patients with single living fetus

  * Patients with gestational or type 2 diabetes
  * Patients on insulin in the 3rd trimester of pregnancy HbA1c level between 7% to 11%
  * All patients require a dating ultrasound to confirm gestational age, viability and rule out multiple.

Exclusion Criteria:

* Patients with type 1 diabetes

  * Patients with congestive heart failure or a history of congestive heart failure
  * Patients with renal insufficiency
  * Patients with intolerance or hypersensitivity to metformin
  * Patients having current significant gastrointestinal problems such as severe vomiting requiring intravenous fluids or hospitalization
  * Presence of acute or chronic metabolic acidosis, including diabetic ketoacidosis, a history of diabetic ketoacidosis or history of lactic acidosis
  * Patients with liver impairment
  * Patients with known higher order pregnancies (twins, triplets, etc.)
  * Patients having a known potentially fetal lethal anomaly

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant women in the 3rd trimester
Enrollment: 150 (Actual)
Dates: Start 2022-07-29 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
Maternal glycemic control 3 months. | 3 months
  blood glucose levels
Maternal insulin requirements | 3 months
  Daily Insulin doses requirements
Maternal Blood glucose readings | 3 months
  fasting and 2 hours post prandial blood sugar.

SECONDARY OUTCOMES:
Maternal weight gain | 3 months
  measured by kilograms
weekly fetal weight gain | 3 months
  measured by ultrasound in grams
increase of attacks of maternal hypoglycemia. | 3 months
  maternal hypoglycemia defined by plasma glucose level below 65 mg/dl
fetal outcomes | 3 months
  intra uterine fetal death (IUFD)
Neonatal outcomes | 1 week
  RDS

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Feig DS, Hwee J, Shah BR, Booth GL, Bierman AS, Lipscombe LL. Trends in incidence of diabetes in pregnancy and serious perinatal outcomes: a large, population-based study in Ontario, Canada, 1996-2010. Diabetes Care. 2014 Jun;37(6):1590-6. doi: 10.2337/dc13-2717. Epub 2014 Apr 4. PMID 24705609
- [Background] Report of the Expert Committee on the Diagnosis and Classification of Diabetes Mellitus. Diabetes Care. 1997 Jul;20(7):1183-97. doi: 10.2337/diacare.20.7.1183. No abstract available. PMID 9203460
- [Background] Ainuddin JA, Karim N, Zaheer S, Ali SS, Hasan AA. Metformin treatment in type 2 diabetes in pregnancy: an active controlled, parallel-group, randomized, open label study in patients with type 2 diabetes in pregnancy. J Diabetes Res. 2015;2015:325851. doi: 10.1155/2015/325851. Epub 2015 Mar 22. PMID 25874236
- [Background] Gibbons A, Flatley C, Kumar S. Cerebroplacental ratio in pregnancies complicated by gestational diabetes mellitus. Ultrasound Obstet Gynecol. 2017 Aug;50(2):200-206. doi: 10.1002/uog.17242. PMID 27549587
- [Background] Langer O. Type 2 diabetes in pregnancy: exposing deceptive appearances. J Matern Fetal Neonatal Med. 2008 Mar;21(3):181-9. doi: 10.1080/14767050801929497. PMID 18297573
- [Background] Lipscombe LL, Hux JE. Trends in diabetes prevalence, incidence, and mortality in Ontario, Canada 1995-2005: a population-based study. Lancet. 2007 Mar 3;369(9563):750-756. doi: 10.1016/S0140-6736(07)60361-4. PMID 17336651
- [Background] Madiraju AK, Erion DM, Rahimi Y, Zhang XM, Braddock DT, Albright RA, Prigaro BJ, Wood JL, Bhanot S, MacDonald MJ, Jurczak MJ, Camporez JP, Lee HY, Cline GW, Samuel VT, Kibbey RG, Shulman GI. Metformin suppresses gluconeogenesis by inhibiting mitochondrial glycerophosphate dehydrogenase. Nature. 2014 Jun 26;510(7506):542-6. doi: 10.1038/nature13270. Epub 2014 May 21. PMID 24847880
- [Background] Murphy HR, Steel SA, Roland JM, Morris D, Ball V, Campbell PJ, Temple RC; East Anglia Study Group for Improving Pregnancy Outcomes in Women with Diabetes (EASIPOD). Obstetric and perinatal outcomes in pregnancies complicated by Type 1 and Type 2 diabetes: influences of glycaemic control, obesity and social disadvantage. Diabet Med. 2011 Sep;28(9):1060-7. doi: 10.1111/j.1464-5491.2011.03333.x. PMID 21843303
- [Background] Salber GJ, Wang YB, Lynch JT, Pasquale KM, Rajan TV, Stevens RG, Grady JJ, Kenny AM. Metformin Use in Practice: Compliance With Guidelines for Patients With Diabetes and Preserved Renal Function. Clin Diabetes. 2017 Jul;35(3):154-161. doi: 10.2337/cd15-0045. PMID 28761217
- [Background] Shobha P, Mathen S, Abraham J. Glycosylated hemoglobin values in nondiabetic pregnant women in the third trimester and adverse fetal outcomes: An observational study. J Family Med Prim Care. 2016 Jul-Sep;5(3):646-651. doi: 10.4103/2249-4863.197313. PMID 28217599